CLINICAL TRIAL: NCT05705960
Title: The Effect of Chestnut Consumption on Modulation of Gut Microbiota and Metabolic Parameters
Brief Title: Chestnut Consumption on Modulation of Gut Microbiota and Metabolic Parameters
Acronym: CULTIVAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Associação Centro de Apoio Tecnológico Agro-Alimentar de Castelo Branco (CATAA) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CULTIVAR
Record Dates: First submitted 2023-01-20; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Diet Habit
Keywords: Chestnut; Gut microbiota diversity; Short chain fatty acid; Lipid
MeSH Terms: conditions — Feeding Behavior | interventions — horse chestnut seed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chestnut (Experimental)
  Interventions: Other: Chestnut

INTERVENTIONS:
Other: Chestnut — Daily consumption of roasted chestnut (150g) for 14 days

SUMMARY:
The chestnut tree (Castanea sativa Mill.) is a species widely cultivated in Portugal, which is a major producer of chestnuts. Nuts are nutritionally interesting, not only because of their content of vitamins, minerals, and phytochemicals but also of their high fiber content.

Fiber, as it is not digested by humans, has a preponderant role in the intestinal microbiota, for its maintenance, and, consequently, has an impact on metabolic status.

The inclusion of foods rich in these components, and with extensive local production, can be an excellent strategy for improving the metabolic parameters of the population.

The main objective of this single group assignment clinical trial is to evaluate the effect of including roasted chestnuts in the daily diet on the composition and diversity of the intestinal microbiota. It is also intended to evaluate metabolic parameters to determine the impact of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian.
* Filling informed consent.
* Body mass index (BMI) between 18,5 kg/m2 and 25 kg/m2.

Exclusion Criteria:

* Chestnut sensibility.
* Chestnut daily consumption in the month before the study initiation.
* Having taken antibiotics within the 6 months prior to beginning the study;
* Use of pro/prebiotics or fiber as a dietary supplement or any food/molecule that modifies intestinal transit time 6 weeks before recruitment.
* Use of laxative 6 weeks before recruitment.
* Specific dietary regimen (e.g., vegan).
* Specific nutritional therapy (e.g. high protein).
* Excessive alcohol consumption.
* Smoking.
* Diagnosis of gastrointestinal pathology, hormonal or thyroid pathology, autoimmune diseases, chronic use of corticosteroids, psychiatric disease or Diabetes Mellitus.
* Use of proton pump inhibitors, antidiabetic drugs, insulin, or statins.
* Pregnant or breastfeeding.
* Participation in another clinical trial within the last 3 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Gut microbiota characterization | 14 days
  Difference in Gut microbiota taxonomic characterization, from baseline to the end of intervention
Changes in Gut microbiota diversity | 14 days
  Difference in Gut microbiota Shannon index, from baseline to the end of intervention

SECONDARY OUTCOMES:
Changes in fasting glucose | 14 days
  Changes in fasting glucose, measured in mg/dL, from baseline to end of intervention
Changes in HOMA-IR | 14 days
  Changes in HOMA-IR from baseline to end of intervention
Changes in total cholesterol | 14 days
  Changes in total cholesterol, measured in mg/dL, from baseline to end of intervention
Changes in LDL cholesterol | 14 days
  Changes in LDL cholesterol, measured in mg/dL, from baseline to end of intervention
Changes in high sensitivity PCR | 14 days
  Changes in high sensitivity PCR, measured in mg/dL, from baseline to end of intervention
Changes in breath H2 | 14 days
  Changes in breath H2, measured in ppm, from baseline to end of intervention
Changes in breath CH4 | 14 days
  Changes in breath CH4, measured in ppm, from baseline to end of intervention
Changes in fecal butyrate | 14 days
  Changes in fecal butyrate, measured in M, from baseline to end of intervention
Changes in fecal acetate | 14 days
  Changes in fecal acetate, measured in M, from baseline to end of intervention
Changes in fecal ALP | 14 days
  Changes in fecal ALP, measured in mg/g feces, from baseline to end of intervention
Changes in fecal LPS | 14 days
  Changes in fecal LPS, measured in EU/mL , from baseline to end of intervention
Changes in IL-1b | 14 days
  Changes in IL1b, measured in pg/mL , from baseline to end of intervention
Changes in TNFa | 14 days
  Changes in TNFa, measured in pg/mL , from baseline to end of intervention
Changes in adiponectin | 14 days
  Changes in adiponectin, measured in ng/mL , from baseline to end of intervention
Changes in leptin | 14 days
  Changes in leptin, measured in ng/mL , from baseline to end of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ana Faria, PhD, Principal Investigator — Universidade Nova de Lisboa
Locations (1):
- Nova Medical School Universidade Nova de Lisboa, Lisbon, Portugal